CLINICAL TRIAL: NCT02043548
Title: Tocilizumab in the Treatment of Refractory Polymyositis and Dermatomyositis
Acronym: TIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chester Oddis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chester Oddis, Chester Oddis, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ML28681
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: dermatomyositis; polymyositis; tocilizumab; Actemra
MeSH Terms: conditions — Dermatomyositis; Polymyositis | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Tocilizumab (Active Comparator): Tocilizumab will be given at a dose of 8mg/kg by IV infusion every 4 weeks at 6 time points (Visits 1, 2, 3, 4, 5 and 6).
  Interventions: Drug: tocilizumab
- Group B: Placebo (Placebo Comparator): Placebo arm - no active drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tocilizumab — given at a dose of 8mg/kg by IV infusion every 4 weeks at 6 time points (Visits 1, 2, 3, 4, 5 and 6).
  Other Names: Actemra
  Arms: Group A: Tocilizumab
Drug: placebo — given by IV infusion every 4 weeks at 6 time points (Visits 1, 2, 3, 4, 5 and 6).
  Arms: Group B: Placebo

SUMMARY:
The purpose of this multi-center pilot study is to determine if the drug tocilizumab (Actemra) is effective in the treatment of patients with refractory adult polymyositis (PM) and dermatomyositis (DM).

DETAILED DESCRIPTION:
Although there are several studies supporting the efficacy of tocilizumab (TCZ) in Rheumatoid Arthritis (RA) and systemic onset juvenile idiopathic arthritis, it's use in other autoimmune disorders has also been propose. A consensus statement on blocking the effects of IL-6 in RA and other autoimmune conditions has been recently published. IL-6 is involved in the growth and differentiation of many inflammatory cells. In addition to its initial role in triggering B-cell stimulating factor, it also induces T cell growth and differentiation and plays a critical role in both adaptive and innate immune responses. IL-6, produced by many cells including T cells, B cells, monocytes and endothelial cells, binds to its receptor (IL-6R) and subsequently triggers several intracellular pathways leading to the release of inflammatory mediators and stimulation of the immune system. Inhibition of IL-6 has been studied in phase II and III clinical trials of RA. It has led to a decrease in acute phase reactants and other indicators of chronic inflammation. IL-6 is also a potential therapeutic target in systemic sclerosis, and since IL-6 induces differentiation of B cells into antibody forming cells and contributes to T cells transforming into effector cells, its use in Systemic Lupus erythematosus (SLE) has also been suggested.

The use of TCZ in myositis proposed in this protocol is supported by the aforementioned rationale and its efficacy in other rheumatologic disorders. Patients with refractory polymyositis (PM) were treated with tocilizumab and responded favorably. In dermatomyositis, tissue inflammation implicates soluble cytokine networks contributing to disease pathogenesis. Work on a mouse model of myositis noted IL-6 as a mediator of muscle inflammation. Other investigators studying peripheral blood samples and clinical data on both adult and juvenile dermatomyositis (DM) noted that serum levels of IL-6 were significantly correlated with disease activity. In this same study, correlations between serum IL-6 levels and both the type I interferon gene and chemokine signatures were also identified in DM. These authors suggest that the coordinated dysregulation of IL-6 production and Type I interferon signaling implicates these pathways as contributing to disease pathogenesis in DM.

In a mouse model of PM, C protein-induced myositis (CIM), the pathology reportedly mimics that seen in human PM. Mice were treated with anti-IL-6 receptor monoclonal antibodies or control antibodies and muscle tissue was histologically and immunohistochemically analyzed. CIM was ameliorated in this mouse model implicating IL-6 in the development of myositis. These results not only identified this model as useful to understanding PM but they suggest that IL-6 blockade be considered as a new therapeutic approach in the treatment of myositis.

Thus, the collective findings described above provide evidence for the involvement of IL-6 in the pathogenesis of both adult PM and DM as well as supporting its role from animal models and human studies.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the trial based on the following criteria:

1. Definite or probable polymyositis (PM )or dermatomyositis (DM) by the criteria of Bohan and Peter (as modified by IMACS) in adults over the age of 18. We will also allow enrollment of juvenile dermatomyositis(JDM) patients (considered to have DM) over the age of 18 who otherwise meet the inclusion criteria stipulated below.
2. Subjects must either have the classic rash(es) of DM (heliotrope, Gottron sign or Gottron papules), possess one of the myositis-associated autoantibodies (e.g. anti-synthetase, anti-signal recognition particle (anti-SRP), anti-Mi-2, anti-PM-Scl, transcription intermediary factor 1-γ (anti TIF1-γ etc.), or have the diagnosis of PM agreed upon by a 3-member Adjudication Committee consisting of a rheumatologist, neurologist and neuromuscular pathologist.
3. Refractory myositis patients are defined (see Section 3.1.1) as having failed (or considered intolerant to) an adequate course of glucocorticoids or having failed glucocorticoids and at least one other immunosuppressive (IS) or immunomodulatory agent (e.g. methotrexate, azathioprine, cyclosporine, tacrolimus, mycophenolate mofetil, cyclophosphamide, Intravenous immunoglobulin (IVIg), anti-tumor necrosis factor (anti-TNF) agents, and rituximab).
4. Subjects with an Manual muscle score (MMT-8) score ≤ 66 (see Appendix B) must also have at least 2 other core set measures meeting the criteria listed below.
5. Subjects with an MMT-8 score > 66 must have at least 3 other core set measures meeting the criteria listed below and a global extramuscular visual analog score (VAS) score on the Myositis Disease Activity Assessment Tool ( MDAAT) ≥ 5cm on a 10cm scale.
6. Criteria for core set measures for study entry:

   1. Patient global VAS with a minimum value of 2.0cm on a 10cm scale.
   2. MD global VAS with a minimum value of 2.0cm on a 10cm scale.
   3. Health Assessment Questionnaire (HAQ) disability index with a minimum value of 0.25
   4. Elevation of at least one of the muscle enzymes (Creatine kinase (CK), aspartate aminotransferase (AST), alanine transaminase (ALT), aldolase, Lactate dehydrogenase (LDH) at a minimum level of 1.3x the upper limit of normal (ULN).
   5. Global extramuscular disease activity score with a minimum value of 1.0cm on a 10cm VAS scale on the Myositis Disease Activity Assessment Tool (MDAAT).
7. If on prednisone, the dose must be stable for 4 weeks prior to the screening visit. Tapering of the prednisone dose will only be allowed after the subject meets the Definition of Improvement (DOI) or if safety/toxicity issues supervene.

   1. Prednisone Tapering: Prednisone should be held constant without tapering or escalation (unless there is a serious adverse event or disease flare) until the subject has achieved the DOI. Then, tapering of prednisone may commence using a schedule approximating a 20-25% taper of the existing dose every 4 weeks based on the clinical judgment of the clinical site investigator. Prednisone tapering using the aforementioned guidelines can be commenced at any time if: (a) the patient achieves the DOI or (b) there are complications or circumstances that, in the clinical site investigator's opinion, necessitate the tapering of corticosteroids.
   2. Prednisone at Entry: It is also recommended that patients be on less than 1mg/kg/day of prednisone at study entry.
   3. Prednisone Dosing During Flare: If in the clinical site investigator's opinion there are complications or worsening of disease that necessitate an increase in the prednisone dose then the smallest reasonable increase should be considered.
8. If an immunosuppressive (IS) agent was discontinued prior to the screening visit there may be a washout as stipulated below or individualized according to the patients treating physician:

   1. 4 week washout for methotrexate
   2. 8 week washout for any other IS agent (e.g. azathioprine, cyclosporine, tacrolimus, mycophenolate mofetil)
   3. 3 month washout for leflunomide, IVIg or cyclophosphamide
   4. 6 month washout for rituximab
   5. 8 week washout for infliximab or adalimumab
   6. 2 week washout for etanercept
   7. 1 week washout for anakinra
9. If an IS agent is continued, the dose must remain stable for 4 weeks prior to enrollment and at least until the DOI is met or if safety/toxicity issues supervene. Concomitant IS medications permitted include methotrexate, azathioprine, cyclosporine, mycophenolate mofetil, and tacrolimus. IVIg will also be allowed as an immunomodulatory agent. Careful patient safety monitoring along with American College of Rheumatology (ACR) guidelines for monitoring these medications will be employed if those toxicity monitoring laboratory studies are not already being assessed as part of this trial. No concomitant biologic agents are allowed (rituximab, anti-TNFs, abatacept) as well as cyclophosphamide or tofacitinib as concomitant immunosuppressive agents. Investigators will be certain to assess and classify adverse events as being secondary to either study drug as well as any concomitant immunosuppressive agent(s). That is, there should be attribution of the adverse event (AE) to the appropriate agent.
10. Normal organ function, except if abnormal due to the disease under investigation
11. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
12. Subject has provided written informed consent.

Exclusion Criteria:

A patient will be excluded if any of the following criteria are met:

1. Subjects under the age of 18.
2. Severe muscle damage defined as a global muscle damage score >5 on a 10cm VAS scale on the Muscle Damage Index (MDI).
3. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 10 years unless related to primary disease under investigation.
4. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
5. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
6. Active tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted.
7. Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
8. Pregnant women or nursing (breast feeding) mothers.
9. Patients with reproductive potential not willing to use an effective method of contraception.
10. History of alcohol, drug or chemical abuse within 1 year prior to screening or any medical condition or physical or psychological state that the PI feels would not allow the subject to safely complete the study.
11. Initiation of an exercise program for muscle strengthening within 4 weeks of the screening visit or initiation of a muscle strengthening exercise program during the study.
12. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
13. Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
14. Previous treatment with the following cell-depleting therapies, including investigational agents or approved therapies: CAMPATH, cluster of differentiation 4 (anti-CD4), cluster of differentiation antigen 5 (anti-CD5), and anti¬CD3.
15. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
16. Previous treatment with tocilizumab (TCZ).
17. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
18. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
19. Patients with lack of peripheral venous access.
20. Body weight of > 150 kg.
21. Abnormal laboratory values noted below:

    1. Serum creatinine > 1.6 mg/dL in female patients and > 1.9 mg/dL in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
    2. Platelet count < (100,000/mm3); hemoglobin < 8.5 g/dl and white blood cell count (WBC) < 3000/mm3; Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3); Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
22. Positive hepatitis B surface antigen or hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester V. Oddis, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - North Shore Long Island Jewish Center, Great Neck, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oddis CV, Reed AM, Aggarwal R, Rider LG, Ascherman DP, Levesque MC, Barohn RJ, Feldman BM, Harris-Love MO, Koontz DC, Fertig N, Kelley SS, Pryber SL, Miller FW, Rockette HE; RIM Study Group. Rituximab in the treatment of refractory adult and juvenile dermatomyositis and adult polymyositis: a randomized, placebo-phase trial. Arthritis Rheum. 2013 Feb;65(2):314-24. doi: 10.1002/art.37754. PMID 23124935
- [Background] Rider LG, Giannini EH, Brunner HI, Ruperto N, James-Newton L, Reed AM, Lachenbruch PA, Miller FW; International Myositis Assessment and Clinical Studies Group. International consensus on preliminary definitions of improvement in adult and juvenile myositis. Arthritis Rheum. 2004 Jul;50(7):2281-90. doi: 10.1002/art.20349. PMID 15248228
- [Background] Kaly L, Rosner I. Tocilizumab - a novel therapy for non-organ-specific autoimmune diseases. Best Pract Res Clin Rheumatol. 2012 Feb;26(1):157-65. doi: 10.1016/j.berh.2012.01.001. PMID 22424201
- [Background] Schoels MM, van der Heijde D, Breedveld FC, Burmester GR, Dougados M, Emery P, Ferraccioli G, Gabay C, Gibofsky A, Gomez-Reino JJ, Jones G, Kvien TK, Murakami M, Nishimoto N, Smolen JS. Blocking the effects of interleukin-6 in rheumatoid arthritis and other inflammatory rheumatic diseases: systematic literature review and meta-analysis informing a consensus statement. Ann Rheum Dis. 2013 Apr;72(4):583-9. doi: 10.1136/annrheumdis-2012-202470. Epub 2012 Nov 10. PMID 23144446
- [Background] Smolen JS, Schoels MM, Nishimoto N, Breedveld FC, Burmester GR, Dougados M, Emery P, Ferraccioli G, Gabay C, Gibofsky A, Gomez-Reino JJ, Jones G, Kvien TK, Murakami M, Betteridge N, Bingham CO 3rd, Bykerk V, Choy EH, Combe B, Cutolo M, Graninger W, Lanas A, Martin-Mola E, Montecucco C, Ostergaard M, Pavelka K, Rubbert-Roth A, Sattar N, Scholte-Voshaar M, Tanaka Y, Trauner M, Valentini G, Winthrop KL, de Wit M, van der Heijde D. Consensus statement on blocking the effects of interleukin-6 and in particular by interleukin-6 receptor inhibition in rheumatoid arthritis and other inflammatory conditions. Ann Rheum Dis. 2013 Apr;72(4):482-92. doi: 10.1136/annrheumdis-2012-202469. Epub 2012 Nov 21. PMID 23172750
- [Background] Muangchan C, Pope JE. Interleukin 6 in systemic sclerosis and potential implications for targeted therapy. J Rheumatol. 2012 Jun;39(6):1120-4. doi: 10.3899/jrheum.111423. Epub 2012 Apr 15. PMID 22505699
- [Background] Shirota Y, Yarboro C, Fischer R, Pham TH, Lipsky P, Illei GG. Impact of anti-interleukin-6 receptor blockade on circulating T and B cell subsets in patients with systemic lupus erythematosus. Ann Rheum Dis. 2013 Jan;72(1):118-28. doi: 10.1136/annrheumdis-2012-201310. Epub 2012 Aug 2. PMID 22858586
- [Background] Narazaki M, Hagihara K, Shima Y, Ogata A, Kishimoto T, Tanaka T. Therapeutic effect of tocilizumab on two patients with polymyositis. Rheumatology (Oxford). 2011 Jul;50(7):1344-6. doi: 10.1093/rheumatology/ker152. Epub 2011 Apr 22. No abstract available. PMID 21515628
- [Background] Scuderi F, Mannella F, Marino M, Provenzano C, Bartoccioni E. IL-6-deficient mice show impaired inflammatory response in a model of myosin-induced experimental myositis. J Neuroimmunol. 2006 Jul;176(1-2):9-15. doi: 10.1016/j.jneuroim.2006.03.026. Epub 2006 May 24. PMID 16725212
- [Background] Bilgic H, Ytterberg SR, Amin S, McNallan KT, Wilson JC, Koeuth T, Ellingson S, Newman B, Bauer JW, Peterson EJ, Baechler EC, Reed AM. Interleukin-6 and type I interferon-regulated genes and chemokines mark disease activity in dermatomyositis. Arthritis Rheum. 2009 Nov;60(11):3436-46. doi: 10.1002/art.24936. PMID 19877033
- [Background] Sugihara T, Sekine C, Nakae T, Kohyama K, Harigai M, Iwakura Y, Matsumoto Y, Miyasaka N, Kohsaka H. A new murine model to define the critical pathologic and therapeutic mediators of polymyositis. Arthritis Rheum. 2007 Apr;56(4):1304-14. doi: 10.1002/art.22521. PMID 17394136
- [Background] Okiyama N, Sugihara T, Iwakura Y, Yokozeki H, Miyasaka N, Kohsaka H. Therapeutic effects of interleukin-6 blockade in a murine model of polymyositis that does not require interleukin-17A. Arthritis Rheum. 2009 Aug;60(8):2505-12. doi: 10.1002/art.24689. PMID 19644888
- [Background] Oddis CV, Rider LG, Reed AM, Ruperto N, Brunner HI, Koneru B, Feldman BM, Giannini EH, Miller FW; International Myositis Assessment and Clinical Studies Group. International consensus guidelines for trials of therapies in the idiopathic inflammatory myopathies. Arthritis Rheum. 2005 Sep;52(9):2607-15. doi: 10.1002/art.21291. No abstract available. PMID 16142757
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult refractory dermatomyositis and polymyositis
Period: Overall Study
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Tocilizumab | Group B: Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 52.3 [31.3 to 83.4] | 50.4 [21.5 to 70.7] | 52.3 [21.5 to 83.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Black or African American | 3 | 3 | 6
  White | 12 | 14 | 26
  Unknown or Not Reported | 2 | 0 | 2
Dermatomyositis vs. polymyositis per treatment group [Count of Participants; unit: Participants]
  Dermatomyositis | 10 | 13 | 23
  Polymyositis | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Compare the Average Total Improvement Scores at Visits 2 Through 7 During the 6-month Treatment Period Between the Treatment and Placebo Arms
Description: The total improvement score was calculated by adding the improvement scores of all six core set measures based on 2016 American College of Rheumatology (ACR)/European League Against Rheumatism(EULAR) myositis response criteria.
  The minimum and maximum values of the average Total Improvement Scores are 0 and 100; The minimum and maximum values of the average Total Improvement Scores of our included patients are 5.0 and 67.1; The higher scores mean a better outcome.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: All participants randomized are included in intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 26.4 (16.8) | 29.3 (16.8)
Statistical Analysis 1: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.86, GEE

2. Secondary Outcome: Comparison of the Time to First Definition of Improvement (DOI) Between the 2 Arms
Description: Time to achieve the first DOI between the treatment and placebo arms.The total improvement score (TIS) is the sum of all 6 improvement scores associated with the change in each core set measure. A TIS >= 20 represents minimal improvement, a score of >=40 represents moderate improvement, and a score of >=60 represents major improvement.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 18 | 18
days | 42.4 [27.5 to 90.4] | 55.5 [29.4 to 114.6]
Statistical Analysis 1: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.77, Log Rank

3. Secondary Outcome: Count of the Adverse Events Between the Treatment and Placebo Arms.
Description: We compared the count of the adverse events between the treatment and placebo arms statistically.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Measure: Number; unit: events
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 18 | 18
events | 14 | 9
Statistical Analysis 1: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.40, binomial test

4. Secondary Outcome: Comparison of the Steroid-sparing Effect (Calculated Using Prednisone Dose Equivalents) Between the Treatment and Placebo Arms
Description: Mean change of steroid dose prednisone equivalent from last visit to baseline visit was compared between the two treatment arms
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: Only 33 of the total 36 patients were included in analysis due to missing data on three participants.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 17 | 16
mg | 0.0 [0 to 0] | 0.0 [0 to 5]
Statistical Analysis 1: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Comparison of Individual Average Core Set Measure in Subjects Over Time Between the 2 Arms (Repeated Measures Analysis)
Description: The core set measure tested was manual muscle testing, and we compared the mean manual muscle test measures in subjects over time.
  The minimum and maximum values of the manual muscle testing are 0 and 150; The minimum and maximum values of the manual muscle testing of our included patients are 97.0 and 150.0; The higher scores mean a better outcome.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 130.7 (16.94) | 137.3 (11.83)
Statistical Analysis 1: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.78, GEE
Statistical Analysis 2: Comparison: Group A: Tocilizumab vs Group B: Placebo; Test type: Superiority; p = 0.19, t-test, 2 sided

6. Secondary Outcome: Magnitude of the Effect Size Between the Both Treatment Arms
Description: Compared the number of subjects meeting total improvement scores >=20 (minimal) and >=40 (moderate) and >=60 (major) based on 2016 ACR EULAR myositis response criteria for treatment group and placebo group. The highest TIS score achieved from week 4 through week 24 was used to determine the effect size between both treatment arms.
Time Frame: Week 4, 8, 12, 16, 20, and 24
Population: The total improvement score was calculated at each timepoint (weeks 4, 8, 12,16, 20 and 24) for each subject. The greatest improvement score achieved for each subject between week 4 through week 24 was reported (minimal, moderate or major improvement).
Measure: Number; unit: participants
Arm/Group | Group A: Tocilizumab | Group B: Placebo
Number analyzed (Participants) | 18 | 18
participants
  Minimal Improvement | 3 | 7
  Moderate Improvement | 4 | 6
  Major Improvement | 3 | 2

ADVERSE EVENTS:
Time Frame: Time frame period beginning with any amount of exposure to Tocilizumab through the protocol-defined follow-up period. Total duration 1 year.
Arm/Group | Group A: Tocilizumab | Group B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 11/18 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Tocilizumab (N=18) | Group B: Placebo (N=18)
Bilateral sub-massive pulmonary embolism (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Tocilizumab (N=18) | Group B: Placebo (N=18)
General disorders and administration site conditions (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Infusion site reaction of swelling, bruising and redness at infusion site.
Sinusitis (Infections and infestations) | 4 (5) | 3 (4)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT02043548/Prot_SAP_000.pdf